CLINICAL TRIAL: NCT05495906
Title: A Study of Reduced Dosing of the Nonavalent HPV Vaccine in Women Living With HIV
Acronym: NOVA-HIV
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Deborah Money, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H22-01707
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: HPV; Human Papilloma Virus; Human Immunodeficiency Virus
Keywords: HPV vaccination
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Routine schedule (Active Comparator): Three doses of 9vHPV vaccine at the routine dosing schedule of 0/2/6 months
  Interventions: Biological: Nonavalent HPV vaccine
- Extended schedule (Experimental): Two doses of 9vHPV vaccine at an expanded dosing schedule of 0/6 months with a third dose given at month 12
  Interventions: Biological: Nonavalent HPV vaccine

INTERVENTIONS:
Biological: Nonavalent HPV vaccine — Routine dosing form and dosage
  Other Names: Gardasil9

SUMMARY:
There are very little data on human papillomavirus (HPV) vaccination among the 18 million women living with HIV (WLWH) globally, who constitute a population most vulnerable to HPV and the resultant cervical cancer. Particularly, there are no data to date on reduced-dose schedules of nonavalent HPV (9vHPV) vaccination in WLWH and there are very little data on the 9vHPV vaccine in this population overall. It is critical to examine the 9vHPV vaccine in WLWH now because the quadrivalent HPV (4vHPV) vaccine has been discontinued. Additionally, in order to reach the World Health Organization's global goal of cervical cancer elimination, we must determine the role of various HPV prevention strategies in this important population including reduced vaccine dosing which can drastically increase the feasibility of HPV vaccination programs globally.

This randomized clinical trial will enrol WLWH aged 18-45 from across Canada who have not previously received an HPV vaccine. Participants will be randomized 1:1 to receive 3 doses of 9vHPV vaccine at the routine vaccine schedule of 0/2/6 months or 2 doses at an expanded schedule of 0/6 months with a third dose at month 12 to adhere to current recommendations for WLWH. We will compare the immune response generated to two versus three doses of 9vHPV vaccine and will follow participants for 2 years to examine the immune response over time.

This study, which builds upon our team's prior work on HPV vaccination in WLWH, will determine whether two doses of 9vHPV vaccine can be used in WLWH instead of three, and will examine additional aspects of HPV vaccination in WLWH including the immune response to three doses, vaccine safety and efficacy, and attitudes towards self-collected HPV samples in this population. These data will inform global public health policy and programming and will inform the global strategy for cervical cancer elimination.

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV
* Has a uterine cervix

Exclusion Criteria:

* Unable to give fully informed consent
* Pregnant or unwilling to avoid pregnancy during vaccination
* Allergy to the vaccine or its components
* Prior receipt of any HPV vaccine

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 275 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Anti-HPV16/18 geometric mean titers (GMTs) at month 7 | Month 7
  Anti-HPV16/18 GMTs at month 7 (1 month post 3rd dose in Group 1 and 1 month post 2nd dose in Group 2)

SECONDARY OUTCOMES:
Anti-HPV16/18 GMTs at month 24 in both groups (i.e. routine and extended interval) | Month 24
Quantitative summarization of survey responses regarding vaccine acceptability, comfort, and willingness to use HPV self-sampling as a screening methodology in future | Month 24

OTHER OUTCOMES:
Anti-HPV6/11/31/33/45/52/58 GMTs at month 7 (1 month post 3rd dose in Group 1 and 1 month post 2nd dose in Group 2) | Month 7
Anti-HPV16/18 GMTs at month 6 (one-dose data) in the extended vaccine schedule group | Month 6
Incidence, type, and severity of 9vHPV significant adverse events in WLWH | Month 24
Incidence rates of abnormal cervical cytology and histology, and breakthrough persistent HPV infection | Month 24
Peak anti-HPV16/18 GMTs to 1 dose at month 1 | Month 1
Viral and bacterial co-infection in the development of cervical dysplasia and vaccine breakthrough HPV infection in WLWH | Month 0-24
Uptake of HPV vaccination in WLWH aged 18-45 across Canada prior to study | Month 0

CONTACTS AND LOCATIONS:
Locations (10):
- Canada (10):
  - Positive Health Services - Fraser Health, Surrey, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier de l'Université Laval, Québec, Quebec
  - Regina General Hospital, Regina, Saskatchewan